CLINICAL TRIAL: NCT06061965
Title: Facilitating Advance Care Planning Discussions Between Patients With Advanced Cancer and Their Family Caregivers Using a Resilience-Building Intervention
Brief Title: Facilitating Advance Care Planning Discussions for People With Advanced Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-0430; K99NR020358-01A1 (NIH)
Record Dates: First submitted 2023-09-25; First posted 2023-09-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-02

CONDITIONS: Resilience, Psychological; Advance Care Planning

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Web-based resilience-building (Experimental): The web-based resilience-building intervention will be implemented on a website and consist of (1) assessments to help participants (a) understand their coping strategies and (b) appraise their beliefs, values, and goals about advance care planning and (2) 6 weekly modules.
  Interventions: Behavioral: Web-based resilience-building intervention

INTERVENTIONS:
Behavioral: Web-based resilience-building intervention — There are 6 modules on the website. Participants will be encouraged to verbalize their impressions of the website prototype.

SUMMARY:
The aims of this study are to (1) identify the advance care planning deliberation process among 20 dyads of patients with advanced cancer and family caregivers and (2) conduct usability testing among 9 dyads to refine the content and design of the web-based resilience-building intervention.

DETAILED DESCRIPTION:
Patients with advanced cancer have not fully benefited from advance care planning due to the high levels of anxiety and depression experienced and other barriers that affect their appraisals and coping. Despite the protective effects of resilience, there have been few clinical trials improving the resilience skills of patients with advanced cancer and their family caregivers to help initiate advance care planning discussions and sustain engagement. This research will provide new insights through using a dyadic intervention approach to advance care planning while developing and evaluating a web-based resilience-building intervention to improve the completion of advance directives, resilience, coping, anxiety, and depression for patients with advanced cancer and their family caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for the study if they (1) are ≥ 18 years of age; (2) have a cancer diagnosis; (3) are able to read and respond to questions in English with minimal assistance from family caregivers for interpretation; (4) have previously completed an advance directive such as a living will; (5) have a family caregiver who serves as a surrogate in the advance directive and is willing to participate in the study; and (6) have access to the internet on a cell phone, laptop, or computer.
* Family caregivers will be eligible if they (1) are ≥ 18 years of age; (2) are able to read and respond to questions in English with minimal assistance from others for interpretation; (3) are identified by the patient as a family caregiver who serves as a surrogate for health care decisions; and (4) have access to the internet on a cell phone, laptop, or computer.

Exclusion Criteria:

* Patients who have cognitive impairment per a Short Portable Mental Status Questionnaire score < 8.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-07-09 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
Usability | Immediately at the end of the usability testing
  Qualitative feedback from participants about the impressions of the website prototype

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States